CLINICAL TRIAL: NCT04698759
Title: Differences in Immune Status and Fecal SCFA Between Indonesian Stunted Children and Children With Normal Nutritional Status
Brief Title: Immune and Scfa Profile of Stunting Children
Status: Completed | Type: Observational
Sponsor: Bina Nusantara University (Other)
Collaborators: Yayasan Rumah Sakit Islam (YARSI) University (Unknown); Universitas Kristen Indonesia (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Ingrid S Surono, Principal Investigator, Bina Nusantara University
Other Study IDs: No.026/VR.RTT/IV/202
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Immune Deficiency; Stunting; Fatty Acid
Keywords: immune status; stunting; Normal Nutritional Status; Indonesian Children; Gut Microbiota; SCFA
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Growth Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample with plasma and serum preparation Fecal sample with DNA extraction Fecal sample with SCFA preparation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stunted subject: Children with stunted status condition based on Z score criteria
  Interventions: Other: No Intervention
- Normal subject: Children with normal status condition based on Z score criteria
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — no Intervention

SUMMARY:
1. Type and Research Design A cross-sectional study design with a quantitative approach will be conducted. Cross-sectional research design is one-time research to find a relationship between the independent variable (risk factor) and the dependent variable (effect).
2. Time and Location of Research The research will be conducted for approximately six months in 2020 at Banten Regency (namely Tegal Ongok and Pasirkarang) and Sumedang Regency.
3. Population and Research Sample The population is children between three and five years old in the village of stunting locus.

The sampling method to be used in this research was quota sampling, namely 50 stunting and 50 healthy children from each Regency.

DETAILED DESCRIPTION:
The variables studied will be the nutritional status of children between three and five years old, the characteristics of these children (age, sex, LBW, birth length, history of immunization, history of diarrhea, history of upper respiratory tract infection, food intake), mother and family characteristics (mother's age, mother's education, mother's occupation, father's occupation), home environment (aspects of the components of the house, aspects of sanitation facilities, aspects of occupant behavior), the composition of the intestinal microbiota. Data will be obtained through measurements, interviews using a questionnaire, and direct observation using a checklist.

Stunting anthropometric measurements are measured based on parameters of length/height according to age compared to the WHO anthropometric standards 2005 and the Indonesian Minister of Health Decree No. 1995 / MENKES / SK / XII / 2010.

The nutritional status of each child included in this study will be quantified using the WHO recommended three nutritional Z-scores namely, height for age (referred to in this study as Zscore

1. weight for age (referred as Z-score
2. and weight for height (referred as Z-score
3. .A structured questionnaire was used for face-to-face interviews with the respective child mother to collect sociodemographic information. In addition, age and anthropometric measurements (height, weight) based on the Department of Health Ministry of Indonesia The regulation will be recorded. For stunting, the thresholds for height-for-age are: 'severely stunted' (<-3 SD); 'stunted' (-3 SD to < -2 SD); 'normal' (-2 SD to +3 SD); 'tall' (> +3 SD). Furthermore, in order to obtain an overall measure of the nutritional status of these children, the children will be classified into weight-for-height categories: 'severely wasted' (<-3 SD); 'wasted' (-3 SD to < -2 SD); 'normal' (-2 SD to +1 SD); 'possible risk of overweight' (+1 SD to +2 SD); 'overweight' (> +2 SD to +3 SD); 'obese' (> +3 SD)

ELIGIBILITY:
Inclusion Criteria:

* Children age : 3 - 5 years old (36-60 months)
* Live in the research area
* Apparently healthy children, after examination by a physician
* Involved in a research study (informed consent signed by parent or guardian)

Exclusion Criteria:

* Children age < 36 month and > 60 month
* Live outside research area
* Unhealthy, after examination by a physician

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: .A cross-sectional study design with a quantitative approach will be conducted. Cross-sectional research design is one-time research to find a relationship between the independent variable (risk factor) and the dependent variable (effect).
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
TGF beta | 1 week analysis
  Unit : pg/mL from serum
sIgA | 1 week analysis
  Unit : ul/ml from feses extract
IL -10 | 1 week analysis
  unit pg/ml from serum
TNF alfa | 1 week analysis
  unit pg/mL from serum
LBP | 1 week analysis
  Unit ul/ml from serum

SECONDARY OUTCOMES:
Short Chain Fatty Acid | 1 months
  Acetate, Propionate, Butyrate, Isobutyric, Isopropionic , unit mM

OTHER OUTCOMES:
Microbiota profile | 2 months
  relative abundance microbiota profile

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid S Surono, PhD, Principal Investigator — Bina Nusantara University
Locations (1):
- University, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grantham-McGregor S, Cheung YB, Cueto S, Glewwe P, Richter L, Strupp B; International Child Development Steering Group. Developmental potential in the first 5 years for children in developing countries. Lancet. 2007 Jan 6;369(9555):60-70. doi: 10.1016/S0140-6736(07)60032-4. PMID 17208643
- [Result] Titaley CR, Ariawan I, Hapsari D, Muasyaroh A, Dibley MJ. Determinants of the Stunting of Children Under Two Years Old in Indonesia: A Multilevel Analysis of the 2013 Indonesia Basic Health Survey. Nutrients. 2019 May 18;11(5):1106. doi: 10.3390/nu11051106. PMID 31109058
- [Derived] Surono IS, Jalal F, Bahri S, Romulo A, Kusumo PD, Manalu E, Yusnita, Venema K. Differences in immune status and fecal SCFA between Indonesian stunted children and children with normal nutritional status. PLoS One. 2021 Jul 29;16(7):e0254300. doi: 10.1371/journal.pone.0254300. eCollection 2021. PMID 34324500